CLINICAL TRIAL: NCT01396174
Title: A Novel Prosocial Online Support Group for Distressed Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Cancer Support Community, Research and Training Institute, Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RCA158877A
Record Dates: First submitted 2011-07-13; First posted 2011-07-18 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; breast tumor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Standard Online Support Group (Active Comparator)
  Interventions: Behavioral: Standard Online Support Group
- Prosocial Online Support Group (Experimental)
  Interventions: Behavioral: prosocial online support group

INTERVENTIONS:
Behavioral: prosocial online support group — Six weekly 1.5 hour online support group meetings facilitated by a Cancer Support Community staff member. This online support group will maximize opportunities to provide help to others.
  Other Names: Life Beyond Cancer
  Arms: Prosocial Online Support Group
Behavioral: Standard Online Support Group — Six weekly 1.5 hour online support group meetings facilitated by a Cancer Support Community staff member. This online support group will focus on encouraging self-expression.
  Other Names: Life Beyond Cancer
  Arms: Standard Online Support Group

SUMMARY:
The investigators hypothesize that breast cancer survivors participating in a prosocial online support group will have a significantly lower mean level of psychological symptoms (anxiety/depression) and higher mean level of sense of purpose post-intervention than participants in a standard online support group.

DETAILED DESCRIPTION:
Psychological distress is a significant problem among breast cancer survivors. Many survivors turn to the internet for information and support, yet few controlled studies have examined the effectiveness and safety of online support groups. The investigators are testing the potential efficacy, acceptability, and feasibility of an innovative theory-based online support group (OSG) for breast cancer survivors. Members of the control group will participate in a standard OSG that encourages self-expression. Members of the experimental condition will participate in a prosocial OSG that provides structured helping opportunities and coaching on how best to give support to others. Participants will complete two telephone interviews and six weekly online support group meetings.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with stage I or II breast cancer in preceding 36 months
* 21-64 years of age
* access to and ability to use a computer and the internet to communicate with others
* fluent in spoken English
* meet the screening criteria for psychological distress (score >7 on either the depression or anxiety subscale of the Hospital Anxiety and Depression Scales

Exclusion Criteria:

* currently taking medication for depression

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | change from baseline to one month post-intervention

SECONDARY OUTCOMES:
Sense of Coherence measure | change from baseline to one month post-intervention
  We are using the Meaningfulness/Purpose in Life subscale of the Sense of Coherence measure to assess sense of purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Lepore, Ph.D., Principal Investigator — Temple University; Joanne Buzaglo, Ph.D., Study Director — Cancer Support Community
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Lepore SJ, Buzaglo JS, Lieberman MA, Golant M, Greener JR, Davey A. Comparing standard versus prosocial internet support groups for patients with breast cancer: a randomized controlled trial of the helper therapy principle. J Clin Oncol. 2014 Dec 20;32(36):4081-6. doi: 10.1200/JCO.2014.57.0093. Epub 2014 Nov 17. PMID 25403218
- [Derived] Lepore SJ, Buzaglo JS, Lieberman MA, Golant M, Davey A. Standard versus prosocial online support groups for distressed breast cancer survivors: a randomized controlled trial. BMC Cancer. 2011 Aug 25;11:379. doi: 10.1186/1471-2407-11-379. PMID 21867502